CLINICAL TRIAL: NCT07013721
Title: A Clinical Study on the Effect of Ultrasound-Guided Transversus Abdominis Plane Block on Postoperative Analgesic Efficacy in Elderly Patients Undergoing Minimally Invasive Gastrointestinal Tumor Surgery
Brief Title: Transversus Abdominis Plane Block on Postoperative Analgesic Efficacy in Elderly Patients Undergoing Minimally Invasive Gastrointestinal Tumor Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director, Department of Anesthesiology (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PLAGH-TAPB-002
Record Dates: First submitted 2025-05-22; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Regional Anaesthesia; Transversus Abdominis Plane Block (TAP Block); Pain, Postoperative
Keywords: Regional Anaesthesia; Transversus abdominis plane block (TAP block); Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — 1,3-bis(4-amidinophenoxy)-2-(4-amidinophenoxymethyl)ethylpropane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transversus abdominis plane block group (Experimental): The procedure was performed by anesthesiologists with extensive expertise in nerve blockade techniques. For upper abdominal surgical incisions, a subcostal approach transversus abdominis plane block (TAPB) was implemented under ultrasound guidance to identify the transversus abdominis plane. A total of 20 mL of 0.33% ropivacaine hydrochloride injection (Naropin®) was incrementally administered, followed by contralateral application using identical techniques, with ultrasonographic confirmation of fusiform drug distribution within the transversus abdominis plane to achieve upper abdominal incision analgesia. For lower abdominal incisions, a lateral approach was employed, with the same dosage of local anesthetic injected at the target site and bilateral blocks performed after confirming fluid dispersion patterns under real-time ultrasound visualization.
  Interventions: Procedure: Transversus Abdominis Plane Block, TAPB
- Non-intervention Control Group (No Intervention)

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block, TAPB — The procedure was performed by anesthesiologists with extensive expertise in nerve blockade techniques. For upper abdominal surgical incisions, a subcostal approach transversus abdominis plane block (TAPB) was implemented under ultrasound guidance to identify the transversus abdominis plane. A total of 20 mL of 0.33% ropivacaine hydrochloride injection (Naropin®) was incrementally administered, followed by contralateral application using identical techniques, with ultrasonographic confirmation of fusiform drug distribution within the transversus abdominis plane to achieve upper abdominal incision analgesia. For lower abdominal incisions, a lateral approach was employed, with the same dosage of local anesthetic injected at the target site and bilateral blocks performed after confirming fluid dispersion patterns under real-time ultrasound visualization.
  Arms: transversus abdominis plane block group

SUMMARY:
Elderly patients undergoing minimally invasive gastrointestinal tumor surgery face complex postoperative pain management due to age-related physiological decline and surgical particularities, where traditional opioids are prone to adverse effects. Our study investigates the clinical analgesic efficacy of ultrasound-guided transversus abdominis plane block (TAPB) in these patients, focusing on analgesic quality, delirium incidence, opioid consumption, and postoperative recovery indicators. This evaluation aims to assess its clinical value and safety while providing evidence-based insights for optimizing perioperative analgesia protocols.

DETAILED DESCRIPTION:
Globally, approximately 30% of surgical patients experience moderate to severe acute postoperative pain annually, with 11% developing severe acute postoperative pain. Inadequate pain control and analgesic administration may precipitate adverse outcomes such as postoperative delirium, a complication particularly prevalent in elderly populations. The concept of multimodal analgesia has emerged to enhance therapeutic efficacy, mitigate adverse effects associated with monotherapy, accelerate postoperative rehabilitation, and improve patient satisfaction. The transversus abdominis plane block constitutes a critical component of multimodal analgesic strategies.

This randomized controlled trial was conducted to compare the differences in postoperative analgesic efficacy between the transversus abdominis plane block intervention group and the non-intervention control group among elderly patients undergoing minimally invasive gastrointestinal tumor surgery. Key evaluation parameters included postoperative pain intensity (assessed via validated pain scales), incidence of postoperative delirium, opioid consumption , and comprehensive postoperative recovery metrics (e.g., length of hospitalization). The study concurrently evaluated the clinical safety profile of transversus abdominis plane block through systematic monitoring of procedure-related complications and adverse events, thereby providing evidence-based data to refine perioperative analgesic protocols and optimize Enhanced Recovery After Surgery (ERAS) pathways in geriatric surgical populations.

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients scheduled for elective minimally invasive gastrointestinal tumor surgery under general anesthesia
2. Age ≥65 years
3. American Society of Anesthesiologists (ASA) physical status classification ≤III
4. Body mass index (BMI) 18-30 kg/m²

Exclusion Criteria:

1. Allergy to anesthetic agents
2. Preoperative chronic pain or chronic use of opioids/nonsteroidal anti-inflammatory drugs (NSAIDs)
3. Contraindications to regional blockade:Local infection at puncture site

   , Coagulopathy (INR >1.5, platelet count <80×10⁹/L)
4. There is cognitive impairment, which is determined based on Mini Mental State Examination (MMSE) scores below the standard threshold
5. Preoperative neurological/psychiatric disorders:Consciousness alterations, Epilepsy, Alzheimer's disease, Parkinson's disease, Schizophrenia, Anxiety or depressive disorders, Hepatic, pulmonary, or renal encephalopathy
6. Recent stroke history
7. Postoperative admission to intensive care unit (ICU)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2026-04-13 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Pain score | 24 hours after surgery
  Pain scores using Numerical Rating Scale (NRS). The Numerical Rating Scale (NRS) assesses pain intensity through patient self-reporting on an 11-point scale ranging from 0 ("no pain") to 10 ("worst pain imaginable"). Patients independently select a single number reflecting their current pain level without clinician interpretation.

SECONDARY OUTCOMES:
pain score | 1, 6, and 48 hours after surgery
  Resting and movement pain scores using Numerical Rating Scale (NRS). The Numerical Rating Scale (NRS) assesses pain intensity through patient self-reporting on an 11-point scale ranging from 0 ("no pain") to 10 ("worst pain imaginable"). Patients independently select a single number reflecting their current pain level without clinician interpretation.
postoperative delirium during hospitalization | Postoperaitve Day 1-5
  The 3D-CAM (3-Minute Diagnostic Interview for CAM-defined Delirium) is a standardized rapid bedside assessment for delirium screening. It evaluates four core features: (1) Acute onset/fluctuating course, (2) Inattention, (3) Disorganized thinking, and (4) Altered level of consciousness. A positive delirium diagnosis requires: Feature 1 AND Feature 2 to be present concurrently, plus at least one of Feature 3 OR Feature 4.
consumption of sufentanil | During the operation
Subjective sleep quality score | The first postoperative day
  Using the scaleRichards-Campbell Sleep Questionnaire (RCSQ) scale. The Richards-Campbell Sleep Questionnaire (RCSQ) is a patient-reported visual analog scale assessing sleep quality in critically ill patients. It evaluates five domains: sleep depth, sleep latency (ease of falling asleep), awakenings (frequency of disruption), sleep efficiency (returning to sleep), and overall sleep quality. Patients mark each item on a 100-mm line (0 = "worst possible" to 100 = "best possible"). The total score is the mean of all domains (range: 0-100), with higher scores indicating better sleep. Administration requires ≤3 minutes and is completed by alert patients upon waking.
the use of a patient-controlled analgesia (PCA) pump | Three days after surgery
length of hospital stay | No more than 4 weeks
Patient satisfaction | From surgery to hospital discharge (up to 4 weeks).
  Postoperative analgesia satisfaction is assessed using an 11-point Numerical Rating Scale (NRS), where 0 = "completely dissatisfied" and 10 = "completely satisfied".
Adverse reactions: Dizziness, nausea and vomiting | Postoperative Day 1-5

IPD SHARING:
Plan to Share IPD: No